CLINICAL TRIAL: NCT07006402
Title: Effects of Reverse Natural Apophyseal Glides as Compared to Ventro-cranial Translatoric Glides in the Management of Upper Thoracic Spine Hypomobility.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/78
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-07

CONDITIONS: Upper Thoracic Spine Hypomobility

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Study Group (A):
  3-4 treatment sessions per week (for 2 weeks)
  1. TENS and Hot pack for 20 minutes.
  2. Reverse NAGs at level T1-T4 In these type of mobilization, the inferior facet glides up on the superior. The mobilizations are repeated <6 times and then movements are reassessed. If no change occurs, the process will be repeated upto 10 minutes with resting period.
  Interventions: Procedure: Reverse NAGS(experimental)
- Control (Active Comparator): Control Group (B):
  3-4 treatment sessions per week (for 2 weeks)
  1. TENS and Hot pack for 20 minutes.
  2. Grade III Ventro-Cranial Translatoric Glides at level T1-T4 The mobilization will be applied and sustained for 30-40 seconds and will be continued for 10-15 minutes in a cyclic manner.
  Interventions: Procedure: Grade III Ventro-Cranial Translatoric Glides(standard protocol)

INTERVENTIONS:
Procedure: Reverse NAGS(experimental) — All participants will receive 2 weeks of intervention with a frequency of 3-4 days/week with a period of rest in between. 20 minutes of TENS+ hot pack will be given followed by Reverse NAGs on hypomobile segments at level T1-T4.
  In these type of mobilization, the inferior facet glides up on the superior. The mobilizations are repeated <6 times and then movements are reassessed. If no change occurs, the process will be repeated upto 10 minutes with resting period.
  Arms: Interventional Group
Procedure: Grade III Ventro-Cranial Translatoric Glides(standard protocol) — All participants will receive 2 weeks of intervention with a frequency of 3-4 days/week with a period of rest in between. 20 minutes of TENS+ hot pack will be given followed by Grade III Ventro-Cranial Translatoric Glides on hypomobile segments at level T1-T4.
  The mobilization will be applied and sustained for 30-40 seconds and will be continued for 10-15 minutes in a cyclic manner.
  The grades of mobilization will be tapered as per individual needs.
  Arms: Control

SUMMARY:
This study is a randomized controlled trial and the purpose of the study is to determine the effects of reverse NAGs as compared to Ventro-cranial Translatoric Glides in upper thoracic spine hypomobility in terms of pain and range of motion.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are :

1. To determine the effects of reverse NAGs as compared to ventrocranial translatoric glide on UPPER BACK PAIN in upper thoracic spine hypomobility.
2. To determine the effects of reverse NAGs as compared to ventrocranial translatoric glide on THORACIC ROM in upper thoracic spine hypomobility.

HYPOTHESIS:

Alternate Hypothesis:

1. There will be a statistically significant difference in the effects of reverse NAGs as compared to ventrocranial translatoric glides in terms of upper back pain in persons with upper thoracic hypo mobility (p<0.05).
2. There will be a statistically significant difference in the effects of reverse NAGs as compared to ventrocranial translatoric glides in terms of thoracic ROM in persons with upper thoracic hypo mobility (p<0.05).

NULL HYPOTHSIS :

1. There will be no statistically significant difference in the effects of reverse NAGs as compared to ventrocranial translatoric glides in terms of upper back pain in persons with upper thoracic hypo mobility (p>0.05).
2. There will be no statistically significant difference in the effects of reverse NAGs as compared to ventrocranial translatoric glides in terms of thoracic ROM in persons with upper thoracic hypo mobility (p>0.05).

RESEARCH DESIGN : Experimental study .Randomized control trail.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both male and females 2. Adults (18-39 years) 3. Upper Thoracic hypomobility (flexion <20° or extension <25° or side bending <20° or rotation <35°)

Exclusion Criteria:

* 1-Ankylosing spondylitis 2-History of Spinal Fusion or spinal surgery (discectomy/laminectomy etc.) 3-Degenerative disc disorders 4-Cervical radiculopathy, Scoliosis 5-Spinal Stenosis or Myelopathy 6-Recent fracture or surgery 7-TB of spine, Spondylolisthesis 8-Not able to attend regular therapy appointments 9-Fibromyalgia/myofascial pain syndrome

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Thoracic Pain | Variable will be assessed at pre and post treatment for the total interval of 2 weeks.
  It will be measured using numeric pain rating scale (NPRS) in which the subjects select a number ranging from 0-10 according to their intensity of pain. '0' score indicates no pain while '10' indicates worst pain experienced.
Range of Motion | Variable will be assessed at pre and post treatment for the total interval of 2 weeks.
  Range of motion will be measured using inclinometer. It will be used to measure range of motion of flexion, extension and lateral flexion on both right and left side on thoracic spine.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan